CLINICAL TRIAL: NCT00019643
Title: Prospective Study of Potential Factors Affecting Weight in Breast Cancer Patients Receiving Adjuvant Chemotherapy
Brief Title: Factors Affecting Weight Gain in Women Receiving Adjuvant Chemotherapy for Breast Cancer
Status: Terminated | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990026; 99-C-0026; NCI-99-C-0020; CDR0000066928; NCT00001796 (obsolete NCT alias)
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2012-03

CONDITIONS: Depression; Stage I Breast Cancer; Stage IIIA Breast Cancer; Nutrition; Stage II Breast Cancer; Psychosocial Effects/Treatment; Quality of Life
Keywords: adult solid tumor; body system/site cancer; breast cancer; cancer; cancer-related problem/condition; depression; depression and suicide; nutrition; psychosocial effects/treatment; quality of life; solid tumor; stage I breast cancer; stage I, II, and IIIA breast cancer; stage II breast cancer; stage III breast cancer; stage IIIA breast cancer; stage IIIB, IV, recurrent, and metastatic breast cancer; stage, breast cancer
MeSH Terms: conditions — Depression; Breast Neoplasms; Neoplasms; Suicide; Recurrence

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
RATIONALE: Chemotherapy may affect various factors that can lead to weight gain.

PURPOSE: Clinical trial to evaluate factors that may affect weight gain in women receiving adjuvant chemotherapy for stage I, stage II, or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the relative contributions of factors that may lead to weight gain in breast cancer patients receiving adjuvant chemotherapy. Factors examined include: Hormonal and growth factor status (follicle stimulating hormone, total, bound, and free estradiol, androgens, sex hormone binding globulin, thyroid hormones, prolactin, insulin-like growth factors I and II, and plasma leptin) Factors affecting energy intake or expenditure (oral intake, physical activity, and resting metabolic rate) Psychological factors (depression and quality of life) II. Evaluate the effect of chemotherapy on hormonal and growth factor status in these patients.

III. Assess the impact of chemotherapy on bone marrow density in these patients.

PROTOCOL OUTLINE:

Data is collected from women diagnosed with primary breast cancer at 3 points (5 visits): (i) after breast cancer surgery, but before chemotherapy begins (2 visits to NIH day hospital 1 week apart); (ii) 2-3 weeks after chemotherapy has ended (2 visits, 1 week apart); and (iii) 6 months after chemotherapy has ended (1 visit). Tests conducted during these visits include evaluation of blood for hormones, growth factors, and leptin; body composition by DXA; visceral and subcutaneous abdominal adipose tissue by an axial CT scan; and evaluation of resting metabolic rate and daily energy expenditure by a single administration of doubly labeled water at visits "a" and "b" during data collection timepoints 1 and 2. Questionnaires assessing epidemiologic risk factors for breast cancer, dietary intake, physical activity, depression, and quality of life are also administered at the three timepoints.

PROJECTED ACCRUAL:

A total of 140 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Histologically proven newly diagnosed stage I, II, or resectable IIIA primary breast cancer Scheduled to receive chemotherapy No distant metastases --Prior/Concurrent Therapy-- Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No concurrent neoadjuvant chemotherapy Endocrine therapy: No concurrent thyroid medication Radiotherapy: No concurrent radiotherapy Surgery: See Disease Characteristics No prior oophorectomy Other: No concurrent alternative medicines alone No concurrent participation in dietary and/or exercise weight loss programs --Patient Characteristics-- Age: 18 to 80 Sex: Female Menopausal status: Premenopausal or postmenopausal Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No physical or mental disability that would preclude completing questionnaires No prior or concurrent diabetes mellitus No prior hypothyroidism or hyperthyroidism

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 1999-08; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noreen Aziz, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Cancer Prevention Studies Branch, Bethesda, Maryland, United States